CLINICAL TRIAL: NCT06543550
Title: Comparison Between the Effects of Implantable Gestrinone and Oral Dienogest in the Treatment of Endometriosis: Randomized Controlled Clinical Trial
Brief Title: Comparison Between the Effects of Implantable Gestrinone and Oral Dienogest in the Treatment of Endometriosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bio Meds Pharmaceutica Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS.001
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Implantable Gestrinone; Dienogest
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implantable Gestrinone (Experimental): Implantation of Gestrinone pellets - Eligible patients will undergo implantation of Gestrinone pellets (bio meds Brasil, Florianópolis, Brazil) subcutaneously, in the gluteal region, using aseptic technique under local anesthesia. Patients will use 1.6mg/kg of weight to treat endometriosis. A second implantation procedure will be performed 6 months after the first, allowing evaluation of the effects of the therapy over a period of 12 months.
  Interventions: Drug: Implantable gestrinone
- Oral Dienogest (Active Comparator): Patients will receive the medication to be administered orally at 2mg daily for 12 months.
  Interventions: Drug: Oral Dienogest

INTERVENTIONS:
Drug: Implantable gestrinone — 1.6mg/kg of weight of gestrinone in pellets (bio meds Brasil, Florianópolis, Brazil) subcutaneously, in the gluteal region.
  Other Names: Gestrinone pellet
  Arms: Implantable Gestrinone
Drug: Oral Dienogest — Administered orally at 2 mg daily
  Arms: Oral Dienogest

SUMMARY:
This study aims to evaluate the effects of therapy with implantable Gestrinone compared to oral Dienogest in relieving complaints related to endometriosis.

DETAILED DESCRIPTION:
Patient recruitment will be carried out on a prospective basis and based on the group of patients from the private Medical Clinics in 4 cities (Campina Grande - Pb, São Paulo - SP, São José dos Campos - SP and Brasilia-DF). The study will include 70 adult female patients of menstrual age, pre-menopause (18 to 45 years old), who seek medical treatment to alleviate complaints related to endometriosis. The selected patients will be randomly allocated into two groups, in a 1:1 ratio. Control Group (n=35) - treatment with oral Dienogest - and Test Group (n=35) - Implantation of Gestrinone pellets. Follow-up visits will be scheduled after 1 week and 1, 3, 6, 9 and 12 months of initiation of therapy. Therapies will be compared with respect to the effects on the severity of dysmenorrhea, dyspareunia and non-cyclical pelvic pain (Verbal Scale and Visual Analogue Scale), level of Uterine Bleeding assessed by PBAC, systemic effects (hormonal, hepatic, lipid profile, cell concentration red, clotting factor - assessed through blood tests), endometriosis lesions, endometrial thickness (transvaginal ultrasound), body composition (bioimpendance test), quality of life (EHP30) and sexual function (female sexual function index ) - FSFI. Data analysis will be carried out using validated statistical software. Chi-square or Fisher's exact tests will be used to compare qualitative variables, while independent t-tests will be used to compare quantitative variables between the two groups. Analysis of variance with repeated measures will be used to compare the average pain intensity over time. The significance level for all tests will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients of menstrual age, pre-menopause (18 to 45 years old), who seek medical treatment to alleviate complaints related to endometriosis, who are not undergoing other therapies to treat them.
* Patients must have a diagnosis of Grade 1 or 2 endometriosis assessed by imaging tests (ultrasound with bowel preparation and/or MRI of the pelvis with bowel preparation)14, have a BMI of up to 25kg/m2, and weigh between 50 and 70kg.

Exclusion Criteria:

* Pregnant patients (supporting test must be presented)
* Breastfeeding women, using other hormonal contraceptive methods or copper or silver IUDs, who have polycystic ovaries, and/or hyperandrogenism.
* Patients using medications that may interfere with androgen metabolism within 4 weeks of screening or during the study.
* Patients with a history of liver disease, cardiovascular disease (myocardial infarction, unstable angina or heart failure), active hepatitis, liver neoplasia or renal failure
* Patient who are scheduled for surgical treatment during the study period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 70 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of dysmenorrhea severity | Pre-treatment, 1 week, 1, 3 , 6 and 12 months
  Patients will be instructed to rate the intensity of dysmenorrhea at each visit after the first month of treatment, using a modified verbal scale from 0 to 3, as suggested by Biberoglu and Behrman. Patients should also rate the intensity of the symptoms using a 100 mm visual analogue scale.
Evaluation of dyspareunia severity | Pre-treatment, 1 week, 1, 3 , 6 and 12 months
  Patients will be instructed to rate the intensity of deep dyspareunia at each visit after the first month of treatment, using a modified verbal scale from 0 to 3, as suggested by Biberoglu and Behrman. Patients should also rate the intensity of the symptoms using a 100 mm visual analogue scale.
Evaluation of non-cyclical pelvic pain severity | Pre-treatment, 1 week, 1, 3 , 6 and 12 months
  Patients will be instructed to rate the intensity of pelvic pain (outside the menstrual period), at each visit after the first month of treatment, using a modified verbal scale from 0 to 3, as suggested by Biberoglu and Behrman. Patients should also rate the intensity of the symptoms using a 100 mm visual analogue scale.
Evaluation of endometriosis foci regression | Pre-treatment, 6 and 12 months
  Assessment of endometriosis lesions and endometrial thickness on Transvaginal Ultrasound with bowel preparation and/or MRI of the pelvis with bowel preparation - All patients will be referred, at pre-treatment and at 6 and 12 month visits, to undergo transvaginal ultrasound to assess the presence or absence of endometriotic lesions, in addition to controlling the thickness of the endometrium.

SECONDARY OUTCOMES:
Evaluation of quality of life | Pre-treatment, 6 and 12 months
  The evaluation of the influence of complaints on the impact of endometriosis on patients' quality of life will be carried out using the EHP-30 questionnaires validated for the Portuguese language.
Evaluation of adverse effect | Pre-treatment, 1 week, 1, 3 , 6 and 12 months
  Evaluation of sings and symptoms. In addition, it will be evaluated at each visit the serum levels of Estradiol, Sex Hormone Binding Globulin (SHBG), Progesterone, Total and free Testosterone, FSH, LH, Hepatic transaminase (TGO, TGP, GGT), Total cholesterol and fractions, Triglycerides, Red cell concentration, Coagulation factors , Homocysteine, Fibrinogen, DHT.
Evaluation of abnormal Uterine Bleeding (AUB) | Pre-treatment, 1, 3 , 6 and 12 months
  The duration and intensity of menstrual flow will be recorded pre-treatment and at each visit after the first month of treatment. Abnormal uterine bleeding will be defined as a PBAC (Pictorial blood loss assessment chart) score greater than 100.
Evaluation of sexual function | Pre-treatment, 1 week, 1, 3 , 6 and 12 months
  The assessment of sexual function (desire, excitement, lubrication, orgasm, satisfaction and pain) will be carried out through the application of the Female Sexual Function Index.
Evaluation of body composition | Pre-treatment, 3 , 6 and 12 months
  Body composition will be assessed using the tetrapolar Bioimpedance test with the Indoby device (weight, percentage of lean mass and fat mass)

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Gm Ignacio Atividade Medica LTDA, Brasília, Federal District
  - Instituto Longevite Servicos Medicos LTDA, Campina Grande, Paraíba
  - Jpml Clinica Medica LTDA, São José dos Campos, São Paulo
  - Dra Juliana Bicca Endocrinologia e Medicina Funcional LTDA, São Paulo

IPD SHARING:
Plan to Share IPD: No
The patients data will be reported together in the final report.